CLINICAL TRIAL: NCT03237923
Title: Evaluation of the EasySense System in Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Memphis (Other)
Responsible Party: Principal Investigator, Sitaramesh Emani, Dr. Sitaramesh Emani, MD, Ohio State University
Other Study IDs: 2016H0069
Record Dates: First submitted 2017-07-18; First posted 2017-08-03 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Congestive Heart Failure
Keywords: fluid
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EasySense device — Implementation of EasySense device during hospitalization and daily post-discharge for thirty days.

SUMMARY:
The EasySense device is a non-invasive device designed to measure lung fluid in patients with Congestive Heart Failure (CHF). This study seeks to evaluate the efficacy of the EasySense system in measuring lung fluid volume.

DETAILED DESCRIPTION:
Across the globe, Congestive Heart Failure (CHF) continues to be the leading cause of mortality and hospitalizations in the 21st century. Despite advancements, prognosis often remains poor and mortality high. Congestive Heart Failure diagnoses are often characterized by frequent hospitalizations and re-admissions, and early detection of pulmonary edema, a chief characteristic of worsening heart failure, may have positive implications in patients' quality of life and frequency of hospitalizations. The EasySense device is a non-invasive device designed to measure lung fluid in patients with CHF. Similar to ultrasound technology, the device uses radiofrequency waves to assess fluid status. The device is placed on the bare skin of the chest and held in place for approximately 60 seconds to obtain a reading.

This study seeks to evaluate the efficacy of the EasySense system in measuring lung fluid volume. Seventy-five patients are sought for enrollment. Patients will be enrolled during their hospital stay, and will be asked to maintain daily EasySense measurements, in addition to other measurements, for thirty days post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Current hospitalization for acute decompensated heart failure requiring IV diuretics or vasoactive drugs
* NYHA class II-IV
* Willing and able to participate in index and follow-up measurements
* Able to speak, read, and write in English
* Knows how to use a smartphone
* Preference for patients who undergo a right heart catheterization or continuous pulmonary artery monitoring upon admission or during hospitalization

Exclusion Criteria:

* Current or planned treatments with any inotropic agents or mechanical support (LVAD, intra-aortic balloon pump, invasive mechanically assisted ventilation) at time of enrollment
* Requiring demand pacing
* Prior heart transplant
* End-stage renal disease on hemodialysis
* Physical deformities in the thorax area that may prevent proper application of EasySense device, as assessed by investigator
* Sign of local rib cage or thoracic lesion or any illness which may be aggravated or cause significant discomfort from application of EasySense device, as assessed by investigator
* Pregnancy or lactation

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study seeks to enroll patients over the age of 21, diagnosed with congestive heart failure, who are admitted to the hospital for acute decompensated heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of volume status to EasySense measurements | 30 days
  Patient volume status extracted from medical records will be compared to what the EasySense device measures.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No